CLINICAL TRIAL: NCT04647864
Title: The Coronary AccEss After Tavi Registry - A Multicenter Prospective Registry for the Coronary Access After TAVI
Acronym: CAvEAT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Padova (Other)
Collaborators: Fondazione GISE Onlus (Other)
Responsible Party: Sponsor
Other Study IDs: CAvEAT
Record Dates: First submitted 2020-11-24; First posted 2020-12-01 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Aortic Valve Disease
MeSH Terms: conditions — Aortic Valve Disease | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (4):
- Group 1: Edwards Sapien 3 and Edwards Sapien 3 Ultra
  Interventions: Device: Transcatheter Aortic Valve Implantation
- Group 2: Medtronic Corevalve Evolut R and Medtronic Corevalve Evolut PRO
  Interventions: Device: Transcatheter Aortic Valve Implantation
- Group 3: Boston Scientific Acurate neo and Boston Scientific Acurate neo2
  Interventions: Device: Transcatheter Aortic Valve Implantation
- Group 4: St. Jude Medical Portico
  Interventions: Device: Transcatheter Aortic Valve Implantation

INTERVENTIONS:
Device: Transcatheter Aortic Valve Implantation — Replacement of the aortic valve of the heart through the blood vessels, delivered via one of several access methods.
  Other Names: Transcatheter Aortic Valve Replacement; Percutaneous aortic valve replacement (PAVR); Percutaneous aortic valve implantation (PAVI)

SUMMARY:
The CAvEAT study is a not for profit, international, multicenter study aimed to assess the feasibility of selective coronary angiography (CA) after Transcatheter Aortic Valve Implantation (TAVI), to investigate predictors of successful selective cannulation (anatomical, technical, etc.) and to investigate if there is a significant difference among different type of transcatheter valves in selective coronary cannulation.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic aortic valve disease (stenosis or combined stenosis and regurgitation) candidate to TAVI according to local Heart Team evaluation, including valve-in-valve procedure due to degeneration of a previously implanted surgical bioprosthesis, who undergo coronary access in the same session of TAVI, immediately after transcatheter valve deployment (the procedures have to be consecutive);
* Provision of signed informed consent;
* Age ≥18 Years.

Exclusion Criteria:

* Chronic Kidney Disease stage IV-V (without dialytic treatment; otherwise, patients in dialytic treatment could be included);
* Current participation in an interventional clinical study;
* Age < 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a symptomatic aortic valve disease (stenosis or combined stenosis and regurgitation), who are candidate to TAVI according to local Heart Team evaluation. Valve-in-valve procedure due to degeneration of a previously implanted surgical bio prosthesis are also included in this study population.
  All consecutive patients who undergo coronary access immediately after TAVI will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-01-28 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Successful selective cannulation of both coronary arteries | Immediately after TAVI
  Successful selective cannulation of both coronary arteries

SECONDARY OUTCOMES:
Successful selective cannulation of only left coronary artery | Immediately after TAVI
  Successful selective cannulation of only left coronary artery (and no cannulation or sub selective cannulation of the contralateral)
Successful selective cannulation of only right coronary artery | Immediately after TAVI
  Successful selective cannulation of only right coronary artery (and no cannulation or sub selective cannulation of the contralateral)

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedale Università Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: Undecided